CLINICAL TRIAL: NCT03707938
Title: BRIGHTSTAR: A Pilot Trial of Local Consolidative Therapy (LCT) With Brigatinib in Tyrosine Kinase Inhibitor-Naive ALK-Rearranged Advanced NSCLC
Brief Title: Local Consolidative Therapy and Brigatinib in Treating Patients With Stage IV or Recurrent Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0598; NCI-2018-02099 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0598 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lung Carcinoma; ALK Gene Rearrangement; Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (brigatinib, LCT) (Experimental): Patients receive brigatinib PO QD on days 1-28. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo LCT for up to 3 weeks in the absence of disease progression or unacceptable toxicity. Within 7 days after completion of LCT, patients receive brigatinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brigatinib; Procedure: Local Consolidation Therapy

INTERVENTIONS:
Drug: Brigatinib — Given PO
  Other Names: Alunbrig; AP 26113; AP-26113; AP26113
Procedure: Local Consolidation Therapy — Undergo local consolidative therapy
  Other Names: LCT; Local Consolidative Therapy

SUMMARY:
This early phase I trial studies the side effects and how well local consolidative therapy (LCT) and brigatinib works in treating patients with non-small cell lung cancer that is stage IV or has come back (recurrent). Giving LCT, such as surgery and/or radiation, after initial treatment may kill any remaining tumor cells. Brigatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving LCT and brigatinib may work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety, tolerability, and feasibility of brigatinib with local consolidative therapy (LCT) in tyrosine kinase inhibitor-naive ALK-rearranged advanced (non-small cell lung cancer) NSCLC.

SECONDARY OBJECTIVES:

I. To determine progression-free survival (PFS) using modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1) in advanced ALK+ NSCLC patients treated with local consolidative therapy (LCT) after achieving stable disease or partial response with first-line brigatinib treatment.

II. To determine overall survival (OS).

III. To assess time to progression (TTP) of non-LCT lesions.

EXPLORATORY OBJECTIVES:

I. To assess time to appearance of new metastatic lesion(s).

II. To determine the utility of pre-treatment, pre-LCT, and post-LCT circulating free tumor deoxyribonucleic acid (DNA) (cfDNA) as a potential prognostic and predictive biomarkers.

II. To evaluate potential impact of LCT on mechanisms of ALK resistance with molecular analysis of post-progression biopsies.

OUTLINE:

Patients receive brigatinib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo LCT for up to 3 weeks in the absence of disease progression or unacceptable toxicity. Within 7 days after completion of LCT, patients receive brigatinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of stage IV NSCLC (or recurrent NSCLC not a candidate for definitive multimodality therapy)
2. Documented ALK re-arrangement as detected by: (1) FISH, (2) IHC, (3) tissue NGS, or (4) cfDNA NGS
3. Subjects can be enrolled as (1) TKI naïve or (2) after ≤ 8 weeks of first-line brigatinib treatment without disease progression.
4. Candidate for local consolidative therapy to at least one site of residual disease
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
6. Males or females aged at least 18 years.
7. Adequate organ function laboratory values, defined as:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L or at least 1500/mm3 or at least 1.5 x 109/L
   2. Platelet count at least 75,000/mm3 or at least 75 x 109/L
   3. Hemoglobin (Hb) at least 9 g/dL (or 5.69 mmol/L) at baseline
   4. Serum creatinine ≤ 1.5 × ULN or ≥ 60 mL/minute for subjects with creatinine levels > 1.5 × the institutional ULN
   5. Serum total bilirubin less than or equal to ≤ 1.5 × ULN or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 × ULN
   6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN except for subjects with liver mets for whom ALT and AST should be ≤ 5× ULN
   7. International Normalized Ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
   8. Activated PTT (aPTT) ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulant
8. Female patients of childbearing potential must have a negative pregnancy test documented at time of screening.
9. Female patients who:

   1. Are postmenopausal for at least 1 year before the screening visit, OR
   2. Are surgically sterile, OR
   3. If they are of childbearing potential, agree to use a highly effective method of contraception from the time of signing the informed consent through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse
10. Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:

    1. Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
    2. Agree to completely abstain from heterosexual intercourse
11. Have normal QT interval on screening ECG evaluation, defined as QT interval corrected (Fridericia) (QTcF) of ≤450 milliseconds (msec) in males or ≤470 msec in females.
12. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

1. Have been diagnosed with another primary malignancy other than NSCLC, except for adequately treated non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or patients with another primary malignancy who are definitively relapse-free with at least 2 years elapsed since the diagnosis of the other primary malignancy.
2. Previously received any prior TKI, including ALK-targeted TKIs. Note: on-going first-line brigatinib use as specified in the Inclusion criteria is allowed.
3. Previously received more than 1 regimen of chemotherapy or immunotherapy for locally advanced or metastatic disease. Note that history of consolidative immunotherapy after concurrent chemoradiotherapy (for locally advanced disease) is allowed.
4. Symptomatic CNS metastasis. Asymptomatic CNS disease requiring increasing dose of corticosteroids within 7 days prior to study enrollment is also not permitted.
5. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Patients with leptomeningeal disease and without cord compression are allowed.
6. The presence of pulmonary interstitial disease, drug-related pneumonitis, or radiation pneumonitis at screening.
7. Have a known or suspected hypersensitivity to brigatinib or its excipients.
8. Have malabsorption syndrome or other gastrointestinal (GI) illness or condition that could affect oral absorption of the study drug.
9. Be pregnant, planning a pregnancy, or breastfeeding.
10. Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

    1. Myocardial infarction (MI) within 6 months prior to the first dose of study drug
    2. Unstable angina within 6 months prior to first dose of study drug
    3. Decompensated congestive heart failure (CHF) within 6 months prior to first dose of study drug
    4. History of clinically significant atrial arrhythmia (including clinically significant bradyarrhythmia), as determined by the treating physician
    5. Any history of ventricular arrhythmia
    6. Cerebrovascular accident or transient ischemic attack within 6 months prior to first dose of study drug
11. Have uncontrolled hypertension. Patients with hypertension should be under treatment on study entry to control blood pressure
12. Have an ongoing or active infection, including, but not limited to, the requirement for intravenous (IV) antibiotics.
13. Have a known history of human immunodeficiency virus (HIV) infection. Testing is not required in the absence of history.
14. Have any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Toxicity data will be summarized using frequency tables. Associations between the types and severity of toxicity and treatment will be evaluated as well.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of brigatinib treatment initiation until disease progression or death, assessed up to 2 years
  The median PFS will be calculated and presented with 2-sided 80% confidence interval (CI). Kaplan-Meier survival probabilities will be plotted over time.
Overall survival (OS) | From the date of brigatinib treatment initiation until date of death from any cause, assessed up to 2 years
  The median OS will be calculated and presented with 2-sided 80% CI. Kaplan-Meier survival probabilities will be plotted over time.
Time to progression of non-local consolidative therapy (LCT) lesion | From the date of brigatinib treatment initiation until progression of a baseline lesion not treated with radiation or surgery, assessed up to 2 years
  The median time to progression of non-LCT lesion will be calculated and presented with 2-sided 80% CI. Kaplan-Meier survival probabilities will be plotted over time.

OTHER OUTCOMES:
Time to appearance of new metastatic lesion(s) (TANM) | From the date of brigatinib treatment initiation until development of a new lesion, assessed up to 2 years
  Descriptive statistics (e.g. median, standard deviations, range) will be used to quantify TANM.
Potential prognostic and predictive biomarkers | Up to 2 years
  Multi-covariate and multivariate analysis tools such as the logistic regression, generalized linear model, classification and regression tree, canonical correlation, correspondence analysis, etc., will be applied to study the association among various immunological markers, genomic markers, treatments, and the toxicity and efficacy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Y Elamin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org